CLINICAL TRIAL: NCT02464150
Title: Gluten Challenge in Celiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other); Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Knut E. A. Lundin, Professor, M.D., PhD., Consultant gastroenterologist, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013/1237
Record Dates: First submitted 2015-03-30; First posted 2015-06-08 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Celiac Disease
Keywords: gluten; antigen-specific T cells; transcriptome
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants are subjected to gluten intervention in an unblinded fashion.
  Interventions: Dietary Supplement: Gluten challenge

INTERVENTIONS:
Dietary Supplement: Gluten challenge — Challenge done in the form of a gluten containing cookie once daily, or up to four slices of regular bread daily.

SUMMARY:
Up till 30 participants with celiac disease on a glutenfree diet are asked to consume gluten containing cookies or bread for 3 days.

Questionnaires and sampling of blood is done before, during and after.

DETAILED DESCRIPTION:
Before and 6 days after start of gluten challenge, blood samples will be collected and analysed by using HLA-tetramers to identify and purify CD4+ gluten-specific T cells by flow cytometry. T cells will undergo transcriptome analysis to get an insight in signalling of antigen-specific cells. Other cell populations like CD8+ T cells and γδ T cells will also be analyzed by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Celiac disease confirmed by biopsy
* Age 18 - 80 years
* Gluten free diet last 6 months
* Subject has received information and signed the informed consent form

Exclusion Criteria:

* Pregnant or breast feeding
* Probability of participant becoming pregnant (f.ex. by not using adequate sexual prevention by woman in fertile age)
* Drugs influencing immune system used last 3 months
* Current infectious disease of moderate or high severity
* Other chronic active intestinal disease
* Serious reaction on small amounts of gluten ingested

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Transcriptome of gluten-specific T cells | Day 6
  Transcriptional differences of glutenspecific vs. unspecific T cells

CONTACTS AND LOCATIONS:
Overall Officials: Knut EA Lundin, MD PhD, Principal Investigator — Oslo University Hospital and University of Oslo
Locations (1):
- Oslo university hospital - Rikshospitalet, Oslo, Norway

REFERENCES:
- [Result] Eggesbo LM, Risnes LF, Neumann RS, Lundin KEA, Christophersen A, Sollid LM. Single-cell TCR sequencing of gut intraepithelial gammadelta T cells reveals a vast and diverse repertoire in celiac disease. Mucosal Immunol. 2020 Mar;13(2):313-321. doi: 10.1038/s41385-019-0222-9. Epub 2019 Nov 14. PMID 31728027
- [Result] Zuhlke S, Risnes LF, Dahal-Koirala S, Christophersen A, Sollid LM, Lundin KE. CD38 expression on gluten-specific T cells is a robust marker of gluten re-exposure in coeliac disease. United European Gastroenterol J. 2019 Dec;7(10):1337-1344. doi: 10.1177/2050640619874183. Epub 2019 Sep 7. PMID 31839959
- [Result] Risnes LF, Eggesbo LM, Zuhlke S, Dahal-Koirala S, Neumann RS, Lundin KEA, Christophersen A, Sollid LM. Circulating CD103+ gammadelta and CD8+ T cells are clonally shared with tissue-resident intraepithelial lymphocytes in celiac disease. Mucosal Immunol. 2021 Jul;14(4):842-851. doi: 10.1038/s41385-021-00385-8. Epub 2021 Mar 2. PMID 33654213
- [Result] Dahal-Koirala S, Risnes LF, Neumann RS, Christophersen A, Lundin KEA, Sandve GK, Qiao SW, Sollid LM. Comprehensive Analysis of CDR3 Sequences in Gluten-Specific T-Cell Receptors Reveals a Dominant R-Motif and Several New Minor Motifs. Front Immunol. 2021 Apr 13;12:639672. doi: 10.3389/fimmu.2021.639672. eCollection 2021. PMID 33927715
- [Result] Christophersen A, Zuhlke S, Lund EG, Snir O, Dahal-Koirala S, Risnes LF, Jahnsen J, Lundin KEA, Sollid LM. Pathogenic T Cells in Celiac Disease Change Phenotype on Gluten Challenge: Implications for T-Cell-Directed Therapies. Adv Sci (Weinh). 2021 Nov;8(21):e2102778. doi: 10.1002/advs.202102778. Epub 2021 Sep 8. PMID 34495570
- [Result] Christophersen A, Zuhlke S, Lund EG, Snir O, Dahal-Koirala S, Risnes LF, Jahnsen J, Lundin KEA, Sollid LM. Pathogenic T Cells in Celiac Disease Change Phenotype on Gluten Challenge: Implications for T-Cell-Directed Therapies. Adv Sci (Weinh). 2022 Dec;9(34):e2205912. doi: 10.1002/advs.202205912. No abstract available. PMID 36482157
- [Result] Stamnaes J, Stray D, Stensland M, Sarna VK, Nyman TA, Lundin KEA, Sollid LM. In Well-Treated Celiac Patients Low-Level Mucosal Inflammation Predicts Response to 14-day Gluten Challenge. Adv Sci (Weinh). 2021 Jan 4;8(4):2003526. doi: 10.1002/advs.202003526. eCollection 2021 Feb. PMID 33643806
- [Result] Tye-Din JA, Skodje GI, Sarna VK, Dzuris JL, Russell AK, Goel G, Wang S, Goldstein KE, Williams LJ, Sollid LM, Lundin KE, Anderson RP. Cytokine release after gluten ingestion differentiates coeliac disease from self-reported gluten sensitivity. United European Gastroenterol J. 2020 Feb;8(1):108-118. doi: 10.1177/2050640619874173. Epub 2019 Sep 3. PMID 32213060
- [Result] Goel G, Tye-Din JA, Qiao SW, Russell AK, Mayassi T, Ciszewski C, Sarna VK, Wang S, Goldstein KE, Dzuris JL, Williams LJ, Xavier RJ, Lundin KEA, Jabri B, Sollid LM, Anderson RP. Cytokine release and gastrointestinal symptoms after gluten challenge in celiac disease. Sci Adv. 2019 Aug 7;5(8):eaaw7756. doi: 10.1126/sciadv.aaw7756. eCollection 2019 Aug. PMID 31457091
- [Result] Risnes LF, Christophersen A, Dahal-Koirala S, Neumann RS, Sandve GK, Sarna VK, Lundin KE, Qiao SW, Sollid LM. Disease-driving CD4+ T cell clonotypes persist for decades in celiac disease. J Clin Invest. 2018 Jun 1;128(6):2642-2650. doi: 10.1172/JCI98819. Epub 2018 May 14. PMID 29757191
- [Result] Dahal-Koirala S, Risnes LF, Christophersen A, Sarna VK, Lundin KE, Sollid LM, Qiao SW. TCR sequencing of single cells reactive to DQ2.5-glia-alpha2 and DQ2.5-glia-omega2 reveals clonal expansion and epitope-specific V-gene usage. Mucosal Immunol. 2016 May;9(3):587-96. doi: 10.1038/mi.2015.147. Epub 2016 Feb 3. PMID 26838051
- [Result] Skodje GI, Sarna VK, Minelle IH, Rolfsen KL, Muir JG, Gibson PR, Veierod MB, Henriksen C, Lundin KEA. Fructan, Rather Than Gluten, Induces Symptoms in Patients With Self-Reported Non-Celiac Gluten Sensitivity. Gastroenterology. 2018 Feb;154(3):529-539.e2. doi: 10.1053/j.gastro.2017.10.040. Epub 2017 Nov 2. PMID 29102613
- [Result] Sarna VK, Skodje GI, Reims HM, Risnes LF, Dahal-Koirala S, Sollid LM, Lundin KEA. HLA-DQ:gluten tetramer test in blood gives better detection of coeliac patients than biopsy after 14-day gluten challenge. Gut. 2018 Sep;67(9):1606-1613. doi: 10.1136/gutjnl-2017-314461. Epub 2017 Aug 4. PMID 28779027
- [Derived] Herfindal AM, Nilsen M, Aspholm TE, Schultz GIG, Valeur J, Rudi K, Thoresen M, Lundin KEA, Henriksen C, Bohn SK. Effects of fructan and gluten on gut microbiota in individuals with self-reported non-celiac gluten/wheat sensitivity-a randomised controlled crossover trial. BMC Med. 2024 Sep 4;22(1):358. doi: 10.1186/s12916-024-03562-1. PMID 39227818